CLINICAL TRIAL: NCT00000440
Title: Sertraline and Naltrexone for Alcohol Dependents
Brief Title: Sertraline and Naltrexone for Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAFAR11222
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-11

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Sertraline

INTERVENTIONS:
Drug: naltrexone (Revia)
Drug: sertraline (Zoloft)

SUMMARY:
This study is a double-blind, placebo-controlled outpatient trial to improve, through the addition of sertraline (Zoloft), the abstinence and relapse rates in alcohol- dependent individuals currently taking naltrexone (Revia).

ELIGIBILITY:
Inclusion Criteria:

* Meets the criteria for alcohol dependence.
* Abstinent from alcohol for a period of at least 5 days and not greater than 30 days.
* Able to read English and complete study evaluations.
* A stable residence and a telephone to ensure that subjects can be located during the study.

Exclusion Criteria:

* Currently meets criteria for substance abuse or dependence with the exception of nicotine dependence.
* Current use of disulfiram (Antabuse) or a MAO Inhibitor.
* Psychotic or otherwise severely psychiatrically disabled (i.e., depressed, suicidal, current mania).
* Major depression at the time of assessment.
* Previous treatment with naltrexone (Revia) for alcohol dependence.
* Significant underlying medical conditions such as cerebral, renal, thyroid, or cardiac disease.
* Abstinent longer than 30 days prior to admission to program.
* Hepatocellular disease or elevated bilirubin levels.
* Females who are pregnant, nursing, or not using a reliable method of birth control.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124
Dates: Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Mount Sinai School of Medicine, New York, New York, United States